CLINICAL TRIAL: NCT02758873
Title: Prescribing Asthma Controller Medication According to Gene Status to Improve Quality of Life in Young People With Asthma
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sussex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14/054/MUK
Record Dates: First submitted 2016-04-20; First posted 2016-05-03 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; montelukast; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personalised Medicine (Experimental): If an add-on controller is required, young people in this arm will be prescribed personalised medicine by results of the genotyping for the adrenergic beta2-receptor gene (ADRB2). Health professional's will be advised to prescribe inhaled salmeterol as 'add-on' controller if trial participants have the Gly/Gly variant on ADRB2, and montelukast if they have Arg/Arg or Arg/Gly variant on ADRB2.
  Interventions: Genetic: Personalised medicine (Salmeterol); Genetic: Personalised medicine (Montelukast)
- Standard care (Active Comparator): If an add-on controller is required, young people will be prescribed medication as per the choice of the primary or secondary care physician, without knowledge of genotypic status.
  Interventions: Other: Standard care

INTERVENTIONS:
Genetic: Personalised medicine (Salmeterol) — If participants require add-on medication and have the Gly/Gly variant on the ADRB2, salmeterol will be prescribed.
  Other Names: Salmeterol
  Arms: Personalised Medicine
Genetic: Personalised medicine (Montelukast) — If participants require add-on medication and have the Arg/Arg or Arg/Gly variant on the ADRB2, montelukast will be prescribed.
  Other Names: Montelukast
  Arms: Personalised Medicine
Other: Standard care — If participants require add-on medication in the arm, they will be prescribed either salmeterol or montelukast according to health professional's choice based on current guidelines.
  Other Names: Salmeterol or montelukast
  Arms: Standard care

SUMMARY:
One in every 11 children in the United Kingdom (UK) has asthma. Children with asthma cough, wheeze and have difficulty breathing. The symptoms which children experience can mean they miss school and makes it difficult for children to take part in playground games and sports. Some have to be admitted to hospital. In fact, in the UK a child is admitted to hospital every 18 minutes because of their asthma.

Effective medicines are available, but a child's response to these medicines is currently unpredictable. This project focuses on an asthma controller medicine called salmeterol. According to reports, tens of thousands of children may be taking this medicine in the UK, but evidence suggests it might not work for around one in seven of them. The study team are investigating whether a new approach to treatment, where prescribing is personalised according to a child's genetic make-up, improves the child's quality of life and provides better control of their asthma. Treatment that is tailored in this way to a person's genetic features is often called 'personalised medicine'.

At the moment, doctors commonly prescribe salmeterol to relieve asthma symptoms if children do not benefit enough from other medicines. But evidence suggests salmeterol may not work properly in children with a certain genetic makeup.

The study team are investigating whether it helps to take children and young people's genetic makeup into account when deciding whether to give them salmeterol or an alternative medicine called montelukast. A simple and inexpensive saliva test can provide the information needed to guide decision making.

DETAILED DESCRIPTION:
Asthma is a common chronic illness in children and young people. It affects, for example, an average of two children in every UK classroom. Initial treatment usually consists of salbutamol used on demand at step 1 of British Thoracic Society (BTS) guidelines. At step 2, regular anti-inflammatory 'controller' therapy starts with the regular use of inhaled corticosteroids such as beclomethasone. Therapeutic efficacy with inhaled steroids usually peaks around 400 micrograms per day of beclomethasone (or equivalent). With inadequate asthma control at step 2, inhaled long-acting β2 agonists (LABA) such as salmeterol, or leukotriene receptor antagonists (LTRA) such as montelukast are added; this represents BTS step 3 for asthma management.

The improvement of asthma-related quality-of-life represents an important goal for the overall pharmacological management of asthma. Juniper has developed and validated questionnaires for the measurement of asthma-related quality-of-life and asthma control in both children and adults. Furthermore, Juniper has defined the minimum improvement in asthma-related quality-of-life that is clinically relevant for participants with this disease. In addition, Juniper has recently validated on-line versions of the asthma-related quality-of-life and asthma control questionnaires in children aged 12 and above. This could provide an opportunity for more long-term and cost-effective comparisons of different asthma treatments through the use of tools that measure asthma control without the need for clinic visits and the completion of paper-based forms.

Overall, in children with asthma managed on step 3, salmeterol appears to provide better asthma control than montelukast in the setting of a randomized controlled trial. However, in real life, the efficacy of salmeterol at step 3 for improving asthma control in individual children appears rather variable, and some children continue to experience day-to-day symptoms and exacerbations.

The investigators showed in a earlier study of 1182 UK children and young adults (4-22 years), 50% of those on regular salmeterol experienced asthma exacerbations over a 6-month period, and 18% required inhaled salbutamol at least daily for symptom relief. A step-wise increase was reported in the risk of asthma attacks related to each copy of the Arg16 allele on the β2 receptor gene (1.7-fold) in asthmatic children and young adults exposed to regular salmeterol in conjunction with inhaled corticosteroids. This led the investigators to hypothesize that, contrary to the observations on the overall population of children and young adults where salmeterol is superior in efficacy to montelukast at step 3, those possessing susceptible Arg16 β2 receptor genotype may experience better asthma control with the addition of montelukast rather than salmeterol as second-line controller medication, in addition to inhaled corticosteroids. As such the investigators elected to identify from their database those children with two copies of the Arg16 polymorphism [i.e. homozygous Arg genotype (∼15% of overall population) who would potentially be at greatest risk]. The mechanism for worse control with regular salmeterol involves a greater susceptibility to agonist-induced down-regulation and uncoupling of airway β2 receptors and associated sub-sensitivity of response in the Arg16 genotype.

The investigators therefore performed a proof-of-concept randomized controlled trial to determine whether genetically susceptible children with homozygous Arg16 genotype experience superior long-term asthma control with montelukast compared with salmeterol when used as tailored second-line controller therapy as add-on to the inhaled steroid fluticasone. The purpose of this preliminary study was to provide evidence to support the potential for personalised medicine based on the individual genotype to improve asthma-related quality-of-life and control. This study was published in 2013, and represents the first prospective randomized controlled study in children with asthma that addresses personalised medicine based on genotype. The results of this study showed that in children expressing the homozygous Arg 16 genotype, in comparison with salmeterol, adding montelukast to inhaled fluticasone significantly improved asthma-related quality-of-life and clinical symptoms, while reducing school absences and inhaled reliever use. The relative benefits of montelukast in comparison with salmeterol became evident within the first 3 months and persisted throughout the whole year.

Subsequently, the investigators systematically searched for other randomised controlled trials comparing the effects of salmeterol (or other long-acting beta2 agonist) with montelukast (or other leukotriene antagonist) within the context of Arg/Gly variation, in children with asthma. No studies could be identified. In particular, there were no trials in either adults or children that have studied quality-of-life, which is a key outcome of interest in the context of asthma-related disability, and which is often unrelated to outcomes such as lung function. The absence of other randomised trials, together with the strength of the investigators proof-of-concept evidence, underscores the need for this powered study.

Rationale:

Children with asthma inadequately controlled on inhaled steroids as 'controller' medication experience greater benefit in asthma-related quality-of-life from allocation of further drug therapy on the basis of their genetic status, in comparison to allocation on the basis of current method of doctor or nurse choice informed by the BTS guidelines.

Primary Objective:

Does the prescribing of asthma controller medication according to beta2 receptor gene status improve quality of life as determined by validated questionnaire (Juniper) in 12-18 year olds with asthma?

Secondary Objectives:

Asthma control, as determined by validated questionnaire 3, 6, 9 and 12 months and an evaluation of how many visits participants report to have attended their General Practitioner (GP) or asthma nurse (non- routine asthma review), A&E or been hospitalised as a result of their asthma . Courses of oral steroids and any other medication taken will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Guardian/Participant is willing and able to provide informed consent/assent
* Physician-diagnosed asthma
* Aged 12-18 years
* Taking inhaled corticosteroids (ICS) with/without second line controller (i.e. LABA/LTRA)

Exclusion Criteria:

* Parent/Guardian/Participant is unwilling or unable to give informed consent/assent
* Known contraindication to montelukast or salmeterol
* Other major airway or lung disease, e.g. chronic lung disease of prematurity, cystic fibrosis, and abnormal airway anatomy
* Pregnant or lactating females (if participants become pregnant during the course of the study they will be asked to inform the research team and be withdrawn from the study)
* Participating in another clinical trial (other than observational trials and registries) concurrently or within 30 days prior to screening for entry into this study
* On step 4 asthma control medication e.g. taking Theophylline, Slo-phylin, Uniphyllin
* Unable to provide saliva/buccal cells for genotyping

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 241 (Actual)
Dates: Start 2016-02; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Asthma Quality of Life Questionnaires with Standardised Activities (AQLQ(S)) | Past two weeks
  A disease-specific health-related quality of life instrument that taps both physical and emotional impact of disease. Participants are asked to think about how they have been during the previous 2 weeks and to respond to each of the 32 questions on a 7-point scale (7 = not bothered at all - 1 = extremely bothered).

SECONDARY OUTCOMES:
Asthma Control Questionnaire (ACQ) | Past week
  The ACQ has 6 questions (the top scoring 5 symptoms, and daily rescue bronchodilator use). Patients are asked to recall how their asthma has been during the previous week and to respond to the symptom and bronchodilator use questions on a 7-point scale (0=no impairment, 6= maximum impairment).
Health care utilisation | 3 months
  Participants will be asked to record how many times they have had to visit their GP or asthma nurse (outside of routine asthma review), A&E or hospital as a result of their asthma over the previous 3 months. Total scores for health care utilisation will be summed over the 12-month study period to create a total score for health care utilisation for each participant. Participants will be asked to enter this data via on the online questionnaire at each 3-month follow up.
Medication use | 3 months
  Participants will be asked to record any courses of oral corticosteroids for asthma and any other medication use over the last 3 months. Medication use (scored by each type of medicinal product) will be summed across the 12 month study period to create total number of additional medicinal product use for each participant. Participants will be asked to enter this data via on the online questionnaire at each 3-month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Somnath Mukhopadhyay, FRCPCH, Principal Investigator — Brighton and Sussex University Hospitals NHS Trust
Locations (5):
- United Kingdom (5):
  - Brighton & Sussex University Hospitals NHS Trust, Brighton, East Sussex
  - Kent, Surrey & Sussex CCGs, Gillingham, Kent
  - NHS Grampian, Aberdeen
  - NHS Tayside, Dundee
  - Bart's Health NHS Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fuhlbrigge AL, Adams RJ, Guilbert TW, Grant E, Lozano P, Janson SL, Martinez F, Weiss KB, Weiss ST. The burden of asthma in the United States: level and distribution are dependent on interpretation of the national asthma education and prevention program guidelines. Am J Respir Crit Care Med. 2002 Oct 15;166(8):1044-9. doi: 10.1164/rccm.2107057. PMID 12379546
- [Background] Juniper EF, Guyatt GH, Ferrie PJ, Griffith LE. Measuring quality of life in asthma. Am Rev Respir Dis. 1993 Apr;147(4):832-8. doi: 10.1164/ajrccm/147.4.832. PMID 8466117
- [Background] Juniper EF, Guyatt GH, Willan A, Griffith LE. Determining a minimal important change in a disease-specific Quality of Life Questionnaire. J Clin Epidemiol. 1994 Jan;47(1):81-7. doi: 10.1016/0895-4356(94)90036-1. PMID 8283197
- [Background] Basu K, Palmer CN, Tavendale R, Lipworth BJ, Mukhopadhyay S. Adrenergic beta(2)-receptor genotype predisposes to exacerbations in steroid-treated asthmatic patients taking frequent albuterol or salmeterol. J Allergy Clin Immunol. 2009 Dec;124(6):1188-94.e3. doi: 10.1016/j.jaci.2009.07.043. PMID 19800676
- [Background] Palmer CN, Lipworth BJ, Lee S, Ismail T, Macgregor DF, Mukhopadhyay S. Arginine-16 beta2 adrenoceptor genotype predisposes to exacerbations in young asthmatics taking regular salmeterol. Thorax. 2006 Nov;61(11):940-4. doi: 10.1136/thx.2006.059386. Epub 2006 Jun 13. PMID 16772309
- [Background] Joos S, Miksch A, Szecsenyi J, Wieseler B, Grouven U, Kaiser T, Schneider A. Montelukast as add-on therapy to inhaled corticosteroids in the treatment of mild to moderate asthma: a systematic review. Thorax. 2008 May;63(5):453-62. doi: 10.1136/thx.2007.081596. PMID 18443162
- [Background] Liggett SB. The pharmacogenetics of beta2-adrenergic receptors: relevance to asthma. J Allergy Clin Immunol. 2000 Feb;105(2 Pt 2):S487-92. doi: 10.1016/s0091-6749(00)90048-4. PMID 10669529
- [Background] Lipworth BJ, Basu K, Donald HP, Tavendale R, Macgregor DF, Ogston SA, Palmer CN, Mukhopadhyay S. Tailored second-line therapy in asthmatic children with the Arg(16) genotype. Clin Sci (Lond). 2013 Apr;124(8):521-8. doi: 10.1042/CS20120528. PMID 23126384
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] British Thoracic Society; Scottish Intercollegiate Guidelines Network. British guideline on the management of asthma. Thorax. 2003 Feb;58 Suppl 1(Suppl 1):i1-94. doi: 10.1136/thorax.58.suppl_1.1i. No abstract available. PMID 12653493
- [Background] Lemanske RF Jr, Mauger DT, Sorkness CA, Jackson DJ, Boehmer SJ, Martinez FD, Strunk RC, Szefler SJ, Zeiger RS, Bacharier LB, Covar RA, Guilbert TW, Larsen G, Morgan WJ, Moss MH, Spahn JD, Taussig LM; Childhood Asthma Research and Education (CARE) Network of the National Heart, Lung, and Blood Institute. Step-up therapy for children with uncontrolled asthma receiving inhaled corticosteroids. N Engl J Med. 2010 Mar 18;362(11):975-85. doi: 10.1056/NEJMoa1001278. Epub 2010 Mar 2. PMID 20197425
- [Background] Juniper EF, Svensson K, Mork AC, Stahl E. Modification of the asthma quality of life questionnaire (standardised) for patients 12 years and older. Health Qual Life Outcomes. 2005 Sep 16;3:58. doi: 10.1186/1477-7525-3-58. PMID 16168050
- [Derived] Ruffles T, Jones CJ, Palmer C, Turner S, Grigg J, Tavendale R, Hogarth F, Rauchhaus P, Pilvinyte K, Hannah R, Smith H, Littleford R, Lipworth B, Mukhopadhyay S. Asthma prescribing according to Arg16Gly beta-2 genotype: a randomised trial in adolescents. Eur Respir J. 2021 Aug 19;58(2):2004107. doi: 10.1183/13993003.04107-2020. Print 2021 Aug. PMID 33479111
- See also: Asthma UK — https://www.asthma.org.uk/advice/resources/#schools